CLINICAL TRIAL: NCT00165204
Title: A Randomized Study of the Effects of Tibolone on Bone Density, Menopause Symptoms and Breast Density in High Risk Women After Prophylactic Oophorectomy
Brief Title: Effects of Tibilone on Bone Density, Menopause Symptoms and Breast Density in Women After Prophylactic Oophorectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other); Massachusetts General Hospital (Other); United States Department of Defense (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 03-363
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: Menopause; Postmenopausal Bone Loss; Breast Cancer
Keywords: Tibolone; High risk women; Oophorectomy; Breast Density; Bone Density
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Breast Neoplasms | interventions — tibolone

INTERVENTIONS:
Drug: Tibolone

SUMMARY:
Women undergoing surgical menopause often experience marked menopausal side effects but are reluctant to use estrogen or other female hormones to ease the transition to menopause because of worries that the hormones may increase breast cancer risks. This study will evaluate tibolone in women experiencing surgical menopause to assess its effects on bone health, menopause symptoms and breast density.

DETAILED DESCRIPTION:
Women interested in participating in this study will be allowed to use hormones to manage symptoms for up to 3 months before beginning the study. Those choosing not to take hormones may enroll in the study immediately.

All women will have a baseline mammogram, breast examination, and bone study density performed, along with blood and urine analysis for measurement of bone markers. They will also be asked to take a questionnaire.

Patients will take either tibolone or placebo once daily for 1 year. Neither the patient or the physician will be aware of which treatment a woman is taking during the study.

Patients will return at 6 and 12 months to have a physical examination, blood work, urine collection and bone studies. At one year, a repeat mammogram will be performed. There are also some questionnaires asking about menopause symptoms that will be performed at intervals during the study.

It is also recommended that patients take calcium and vitamin D throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Good overall health
* Premenopausal at the time of enrollment if before their oophorectomy
* Will undergo or have undergone an oophorectomy
* Negative breast examination and negative breast imaging studies

Exclusion Criteria:

* History of breast cancer, ductal carcinoma in situ (DCIS) or other cancer except for carcinoma in situ of the cervix or basal cell carcinoma of the skin
* History of ovarian cancer, breast cancer (or DCIS) or other malignancy
* Low bone mass compared with age-adjusted controls
* Current or recent exposure (within 3 months) to medications that alter bone metabolism
* Estrogens, progesterones, androgens, tamoxifen or raloxifene within 3 months of randomization
* History of significant medical problems potentially related to estrogens
* History of Paget's disease of bone, ankylosing spondylitis, rheumatoid arthritis or other metabolic bone disease, vitamin D deficiency, hyperparathyroidism, or newly diagnosed hyperthyroidism
* Body mass index (BMI) > 32
* High-density lipoprotein (HDL) cholesterol < 40 mg/dl
* Women whose uterus was retained and who have a history of uterine abnormalities

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2004-04; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
To compare bone mineral density and markers of bone turnover following oophorectomy in patients receiving tibolone versus placebo

SECONDARY OUTCOMES:
To compare changes in menopausal symptoms and mammographic breast density in women taking tibolone to women taking placebo

CONTACTS AND LOCATIONS:
Overall Officials: Judy Garber, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

REFERENCES:
- [Derived] McCauley LS, Ghatas MP, Sumrell RM, Cirnigliaro CM, Kirshblum SC, Bauman WA, Gorgey AS. Measurement of Visceral Adipose Tissue in Persons With Spinal Cord Injury by Magnetic Resonance Imaging and Dual X-Ray Absorptiometry: Generation and Application of a Predictive Equation. J Clin Densitom. 2020 Jan-Mar;23(1):63-72. doi: 10.1016/j.jocd.2018.12.003. Epub 2018 Dec 15. PMID 30638769